CLINICAL TRIAL: NCT06324266
Title: Study on the Efficacy and Safety of Low-dose Cyclophosphamide as Maintenance Therapy for Multiple Myeloma Unsuitable for Transplantation
Brief Title: Study on the Efficacy and Safety of Low-dose CTX as Maintenance Therapy for MM Unsuitable for Transplantation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Feng Li, Clinical Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023NZKY-044-02
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — Cyclophosphamide; Lenalidomide; vicilin protein, plant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm CTX (Experimental): Cyclophosphamide monotherapy: CTX, 0.1g×7days，1/every other week, 28 days per course of treatment,total two years
  Interventions: Drug: Cyclophosphamide
- arm Len (Placebo Comparator): Lenalidomide monotherapy:Len,10mg/day×21days， 28 days per course of treatment,total two years
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Cyclophosphamide — Standard risk group MM patients who achieve VGPR or above after initial induction and consolidation therapy and are not suitable transplantation, are maintained with Cyclophosphamide monotherapy for 2 years.
  Other Names: CTX
  Arms: arm CTX
Drug: Lenalidomide — Standard risk group MM patients who achieve VGPR or above after initial induction and consolidation therapy and are not suitable transplantation, are maintained with Lenalidomide monotherapy for 2 years.
  Other Names: Len
  Arms: arm Len

SUMMARY:
The investigators will conduct randomized and controlled clinical studies in order to preliminarily explore the efficacy and safety of low-dose cyclophosphamide and lenalidomide in maintenance therapy for MM that is not suitable for transplantation in the standard-risk group.

DETAILED DESCRIPTION:
The investigators will conduct randomized and controlled clinical studies to preliminarily explore the efficacy and safety of low-dose cyclophosphamide in maintenance therapy for MM that is not suitable for transplantation in the standard -risk group. Standard risk group MM patients who achieve VGPR or above after initial induction and consolidation therapy will use cyclophosphamide or lenalidomide as maintain therapy for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. After induction and consolidation therapy (8 courses of chemotherapy), MM patients in the standard-risk group who were initially unsuitable for transplantation achieved a therapeutic effect of VGPR or above;
2. Secretory MM with measurable indicators;
3. Age ≥ 18 years old, gender unlimited;
4. No obvious dysfunction of heart, lungs, etc. (≤ Grade I);
5. General KPS ≥ 70% (excluding those caused by pathological fractures and bone pain).

Exclusion Criteria:

1. Cytogenetic high-risk patients;
2. Recurrent or refractory MM;
3. Using autologous hematopoietic stem cell transplantation as a consolidation therapy;
4. The therapeutic effect did not reach VGPR or above before enrollment;
5. Asymptomatic MM;
6. No measurable indicators;
7. KPS<50%(excluding those caused by pathological fractures）；
8. Dysfunction of heart, lungs, etc. (> Grade I);
9. Unable to cooperate in observing adverse reactions and therapeutic effects;
10. Pregnancy, breastfeeding, or refusal of contraception by women;
11. There is drug abuse and medical, psychological, or social conditions that may interfere with patients participating in research or evaluating research results;
12. Any unstable or potentially endangering patient safety and compliance with the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS1 | 3 years
  Progression-free Survival 1

SECONDARY OUTCOMES:
Incidence of Efficacy as assessed by IMWG | 3 years
  Efficacy assessed by IMWG
Incidence of Safety as assessed by CTCAE 4.0 | 3 years
  Safety assessed by CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Li Feng, Doctor, Principal Investigator — Department of Hematology of Jinling Hospital
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No